CLINICAL TRIAL: NCT04952142
Title: Minimal Water Exchange Versus Left Water Exchange in Unsedated Colonoscopy: a Randomized Controlled Trial.
Brief Title: Minimal Water Exchange Versus Left Water Exchange in Unsedated Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021CR320
Record Dates: First submitted 2021-06-18; First posted 2021-07-07 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-04

CONDITIONS: Water Exchange Colonoscopy
Keywords: water-aided colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimal water exchange (Experimental): We suctioned the lumen and infused water by constant pressure on the air-water valve button of the endoscope at the rectum to open the lumen.
  Interventions: Other: minimal water exchange
- traditional water exchange colonoscopy (No Intervention): The water exchange colonoscopy reached the cecum through continuous infusion and suction of water in the whole colon via an additional flushing pump.

INTERVENTIONS:
Other: minimal water exchange — Use a new technique, minimal water exchange colonoscopy, which adds the infusion of modest amounts of water by constant pressure on the air-water valve button of the endoscope to achieve intubation.
  Arms: minimal water exchange

SUMMARY:
Minimal water exchange colonoscopy is theoretically more convenient and faster than water exchange colonoscopy. But few studies compared the differences between the two methods. Therefore, we attempted to evaluate the effect of minimal water exchange colonoscopy prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years for unsedated colonoscopy for colorectal cancer screening, polyp surveillance, or polyp resection were enrolled.

Exclusion Criteria:

* Patients who underwent sedation or analgesia before colonoscopy, and were reluctant to cooperate or provide informed consent. Those who were suffering from too serious diseases to tolerate the examination. The intestinal segment was incomplete or the colonoscopy did not reach the cecum.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
VRS-4 pain scores | 30 minutes.
  a 4-point verbal rating scale (VRS-4) with self-explanatory categories (no, slight, moderate, or severe pain).

SECONDARY OUTCOMES:
Adenoma detection rate. | 40 minutes.
  The proportion of patients in whom at least one adenoma is detected.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We might share our data when all related studies are published, E-mails could be sent to: cenqliu@163.com.